CLINICAL TRIAL: NCT00502801
Title: A Phase 2 Study of Doripenem In The Treatment of Nosocomial and Ventilator-Associated Pneumonia In Hospitals
Brief Title: An Effectiveness, Safety, and Microbiology Study of Doripenem in Patients With Nosocomial (Hospital-acquired) Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012931; DORIINI2002 (Other: PriCara, Unit of Ortho-McNeil, Inc.)
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Pneumonia; Bacterial Pneumonia; Ventilator-Associated Pneumonia; Infections, Nosocomial
Keywords: Pneumonia; Lung Infection; Bacterial Infection; Hospital-Acquired Infection; Ventilator Infection; Antibiotic Therapy
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial; Pneumonia, Ventilator-Associated; Cross Infection; Bacterial Infections | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doripenem (Experimental): 1g i.v. infused over 4 hours every 8 hours for 8 to 14 days
  Interventions: Drug: doripenem

INTERVENTIONS:
Drug: doripenem — 1g i.v. infused over 4 hours every 8 hours for 8 to 14 days

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of doripenem monohydrate in the treatment of patients with nosocomial (hospital-acquired) pneumonia.

DETAILED DESCRIPTION:
Nosocomial pneumonia (NP) accounts for approximately 15% of all hospital-acquired infections. The incidence of NP rises in patients who are on breathing machines. The death rate for NP can be as high as 30%. NP caused by bacteria, such as Pseudomonas aeruginosa, has been associated with an increased death rate compared to other pathogens. Prompt use of appropriate antibiotics is essential. Compounding the issue of nosocomial infections is the increasing rate to which bacteria develop resistance to antibiotics. This hospital based trial is studying doripenem in patients who have nosocomial pneumonia to see if it is effective against bacteria associated with this serious bacterial infection. The duration of treatment can be anywhere from 8 to 14 days. Safety evaluations, such as vital signs and laboratory tests will be performed upon enrollment, after 4 days on therapy, after 9 days on therapy for those on greater than 8 days, at the end of therapy, 7 to 14 days after the end of therapy, and 28 to 35 days after the end of therapy. Adverse events will be collected throughout the study. Clinical response to doripenem therapy will be assessed 7 to 14 days after the end of therapy and the long-term clinical response to doripenem therapy will be assessed 28 to 35 days after the end of therapy. Doripenem IV will be administered for a duration of treatment from 8 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Nosocomial Pneumonia or Ventilator-Associated Pneumonia
* All patients must be hospitalized throughout the treatment period
* Patients must have microbiological samples (respiratory secretions) suitable for culture and microscopy

Exclusion Criteria:

* Known or suspected severe kidney impairment
* Known or suspected liver dysfunction
* Treatment with any investigational drug or device within 30 days before enrollment
* Patients with one or more of the following: cystic fibrosis, lung abscess, active tuberculosis
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PriCara, Unit of Ortho-McNeil, Inc. Clinical Trial, Study Director — PriCara, Unit of Ortho-McNeil, Inc.
Locations (40):
- United States (24):
  - Palm Springs, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Hazard, Kentucky
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Grand Rapids, Michigan
  - Columbia, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Buffalo, New York
  - Flushing, New York
  - Jamaica, New York
  - Toledo, Ohio
  - Providence, Rhode Island
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Norfolk, Virginia
  - Morgantown, West Virginia
- Argentina (2):
  - Buenos Aires
  - Santa Fe
- Canada (2):
  - Oshawa, Ontario
  - Chicoutimi, Quebec
- Concepción, Chile
- Croatia (2):
  - Avenija Gojka Suska 6
  - Zagreb
- Argenteuil 95 95, France
- India (5):
  - Jaipur
  - Kozhikode
  - Manipal
  - Noida
  - Pune
- Novosibirsk, Russia
- Ukraine (2):
  - Kharkiv
  - Ukraine Poltava

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two enrolled subjects didn't take study medication and weren't qualified for safety population.
Groups:
- Doripenem: 1g i.v. infused over 4 hours every 8 hours from day 1 to day 8 to 14, depending on length of treatment
Period: Treatment Period
Arm/Group | Doripenem
Started | 183
Completed | 129
Not Completed | 54
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 7
Not completed — Death | 14
Not completed — OTHER | 30
Period: End of Therapy to Test of Cure
Arm/Group | Doripenem
Started | 129
Completed | 121
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Death | 3
Not completed — OTHER | 2

BASELINE CHARACTERISTICS:
Arm/Group | Doripenem
Number analyzed (Participants) | 183
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (20.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 112
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 4
  CANADA | 6
  CHILE | 9
  CROATIA | 21
  FRANCE | 6
  INDIA | 10
  RUSSIA | 2
  UKRAINE | 5
  USA | 120
race [Number; unit: participants]
  AMERICAN INDIAN OR ALASKA | 2
  ASIAN | 14
  BLACK OR AFRICAN AMERICAN | 14
  OTHER, SPECIFY | 2
  WHITE | 151
ethnicity [Number; unit: participants]
  HISPANIC OR LATINO | 20
  NOT HISPANIC OR LATINO | 158
  OTHER | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (8.63)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rates and 95% Confidence Intervals at the Test-of-Cure Assessment.
Description: The table below shows the percentage of subjects who had a clinical response of "clinical cure" at the Late Follow-up Visit as assigned by the medical monitor. A clinical response of "clinical cure" is defined as no further antibacterial therapy needed for treatment of the infection.
Time Frame: 5 to 21 days after the last dose of study therapy, or at early termination.
Population: Clinically Evaluable: Subset of the ITT population who received at least 5 days of study medication unless deemed a clinical failure with at least 2 full days of therapy, and excluding those subjects with a clinical outcome of Not Evaluable at the TOC assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doripenem
Number analyzed (Participants) | 122
Percentage of participants
  All Clinically Evaluable Subjects | 63.9 [54.7 to 72.4]
  Subjects with Nosocomial Pneumonia | 66.0 [51.7 to 78.5]
  Subjects with Ventilator Associated Pneumonia | 64.4 [50.9 to 76.4]
  Subjects with Healthcare Associated Pneumonia | 50.0 [18.7 to 81.3]

2. Secondary Outcome: Clinical Response Rates at the Late Follow-up Assessment.
Description: as for outcome 1
Time Frame: 28 to 35 days after last dose of study therapy
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Doripenem
Number analyzed (Participants) | 78
Percentage of participants
  All Clinically Evaluable Subjects | 83.3
  Subjects with Nosocomial Pneumonia | 82.9
  Subjects with Ventilator Associated Pneumonia | 84.2
  Subjects with Healthcare Associated Pneumonia | 80.0

ADVERSE EVENTS:
Arm/Group | Doripenem
Serious Adverse Events (participants affected / at risk) | 70/183
Other Adverse Events (participants affected / at risk) | 93/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=183)
Neutropenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 6
Cardiac Failure Congestive (Cardiac disorders) | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 6
Cardiopulmonary Failure (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 1
Sickle Cell Anaemia (Congenital, familial and genetic disorders) | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 1
Pancreatic Fistula (Gastrointestinal disorders) | 1
Multi-Organ Failure (General disorders) | 1
Ulcer (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Lung Infection Pseudomonal (Infections and infestations) | 1
Meningitis Bacterial (Infections and infestations) | 1
Meningoencephalitis Herpetic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Postoperative Wound Infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Renal Abscess (Infections and infestations) | 1
Retroperitoneal Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Septic Shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Feeding Tube Complication (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 2
Weaning Failure (Injury, poisoning and procedural complications) | 1
White Blood Cell Count Increased (Investigations) | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anoxic Encephalopathy (Nervous system disorders) | 1
Cerebral Ischaemia (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Psychomotor Hyperactivity (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Obstructive Uropathy (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Renal Failure Acute (Renal and urinary disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9
Rash Papular (Skin and subcutaneous tissue disorders) | 1
Air Embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=183)
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocythaemia (Blood and lymphatic system disorders) | 11
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 10
Pyrexia (General disorders) | 12
Fungal Infection (Infections and infestations) | 17
Urinary Tract Infection (Infections and infestations) | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 21
Hypertension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days